CLINICAL TRIAL: NCT06774365
Title: CARdiac Imaging and BIomarkers in the Diagnosis of Antibody Mediated Rejection in Heart Transplantation
Acronym: CARIBIAM
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: CARIBIAM; PNRR-MCNT2-2023-12377618 (Other Grant/Funding Number: Ministero della salute)
Record Dates: First submitted 2025-01-09; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Heart Transplantation; Rejection Heart Transplant; HLA Antigens

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EDTA blood samples, from which cfDNA will be extracted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of thisobservational study is to systematically assess the presence and distribution of CMR-defined inflammation and fibrosis in clinically stable HT recipients with DSA detected during active screening for AMR surveillance. The main outcome is to study the prevalence of fibrosis, edema and of altered T1 mapping values in patients with DSA and the prevalence of patients with DSA among all the enrolled patients

DETAILED DESCRIPTION:
This is a multicentric prospective study with experimental sample collection. Therapy and procedures will be performed according to clinical practice and current guidelines. Caring physicians will be blinded to the results of study specific assays, which will not be used to change standard cynical decision making. Patients will be enrolled in the study at the time of the DSA assay performed in the context of standard surveillance (yearly monitoring for anti-HLA antibodies is recommended by current guidelines and is part of routine clinical practice). At study entry patients will receive blood sampling to assay dd-cfDNA (centralized laboratory) and T-reg populations (local laboratory). Clinical characteristics, medical history, and results of standard laboratory tests will be collected at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years

  * Post heart transplantation follow-up between 1 and 15 y
  * Ambulatory clinical stable
  * Left ventricular ejection fraction (LVEF) > 40% (as assessed by complete cardiac ultrasound within 3 months before the enrolment)

Exclusion Criteria:

* Unplanned hospitalization for cardiovascular causes in the previous three months

  * Biopsy-proven cellular (2R or greater) or AMR (pAMR> 1 ) in the previous 3 months
  * Any contraindication to CMR
  * Known pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinically stable adult heart transplanted patients will be consecutively enrolled during the routinely outpatient evaluation in the participating centers after IRB approval.
  Heart Failure and Transplant Unit of IRCCS AOUBO will be the project leader and coordinate the overall study. We plan a one year period for the enrollment and eight months for the follow-up.
  Patients will be treated and followed according to the routinary clinical practice of each participating center.
Sampling Method: Non-Probability Sample
Enrollment: 683 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
prevalence of fibrosis, edema and of altered T1 mapping values in patients with DSA | 5 years
  prevalence
prevalence of patients with DSA among all the enrolled patients | 5 years
  prevalence

SECONDARY OUTCOMES:
differences in dd-cfDNA in patients with and without DSA | 5 years
  differences in dd-cfDNA
differences in T-reg subpopulation in patients with and without DSA | 5 years
  differences in T-reg subpopulation
differences in T-reg and dd-cfDNA in patients with and without abnormal CMR | 5 years
  differences in T-reg and dd-cfDNA
change in DSA, biomarkers and CMR findings after vs before AMR treatment | 5 years
  change in DSA
MACE occurrence | 5 years
  MACE occurrence

CONTACTS AND LOCATIONS:
Overall Officials: Luciano Potena, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy